CLINICAL TRIAL: NCT01460394
Title: Establishment of Normative Data of Brain Network Activation (BNA) Using Evoked Response Potentials in Adolescents and Young Adults
Brief Title: Normative Data of Brain Network Activation in Adolescents and Young Adults
Status: Completed | Type: Observational
Sponsor: ElMindA Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: ELM-02
Record Dates: First submitted 2011-10-16; First posted 2011-10-26 (Estimated); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Healthy Controls
Keywords: Healthy; Control

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy adolescents and young adults

SUMMARY:
Establish normative data of ElMindA's Brain Network Activation (BNA) using evoked response in two age groups: adolescents and young adults.

DETAILED DESCRIPTION:
Currently, there is no reliable, practical, and non-invasive method for assessing changes in electrophysiological activity of the brain associated with brain-related pathologies, e.g., concussion, ADHD, autistic spectrum disorders (ASD), etc. Event Related Potentials (ERPs), which are temporal reflections of the neural mass electrical activity of cells in specific regions of the brain that occur in response to stimuli, may offer such a method, as they provide both a noninvasive and portable measure of brain function. The ERPs provide excellent temporal information, but spatial resolution for ERPs has traditionally been limited. However, by using high-density electroencephalograph (EEG) recording spatial resolution for ERPs is improved significantly. The paradigm for the current study will combine neurophysiological knowledge with mathematical signal processing and pattern recognition methods (BNA) to temporally and spatially map brain function, connectivity and synchronization.

The need of objective measures that will help the clinician in its decision making in brain-related pathologies is recognized. BNA is a new imaging modality that has been developed to fill this gap.

ELIGIBILITY:
Inclusion Criteria:

* Age 15-24 years.
* Willingness to participate and able to give informed assent (child) and/or consent (parent for minors or adult 18+ years of age for self).

Exclusion Criteria:

* Currently participate in a contact sport (e.g., football, hockey, soccer, rugby, lacrosse, martial arts).
* Currently with lice, open wounds on scalp.
* Any chronic disease.
* Any psychiatric disorder, e.g., depression, bipolar disorder, schizophrenic disorder, etc.
* Any CNS neurologic disorder, e.g., epilepsy, seizures, etc.
* Any neuropsychological disorders, e.g.: ADHD, Autistic Spectrum Disorder (ASD), etc.
* History of Special education, e.g., reading disorder (dyslexia), writing disorder (dysgraphia), math disorder (dyscalculia), nonverbal learning disorder.
* History of any medication affecting CNS within the last 3 months, e.g., antidepressants, anticonvulsants, psychostimulants, first generation antihistamines, etc.
* Substance abuse in the last 3 months.
* Significant sensory deficits, e.g., deafness or blindness.
* History of any brain trauma.

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Experimental subjects will include males and females recruited from the Kansas City metropolitan area, Vince & Associates Clinical Research's database and from referrals.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2011-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Functional networks of brain activity in healthy individuals measured using analysis of EEG Event Related Potential (ERP) data | 1 week
  The study outcome measure are functional networks of brain activity of healthy adolescents (age 15-18 years) and young adults (19-24 years) established based on an analysis of EEG data recorded while study subjects perform ERP tasks

CONTACTS AND LOCATIONS:
Overall Officials: Bradley D. Vince, D.O., Principal Investigator — Vince and Associates Clinical Research
Locations (1):
- Vince and Associates Clinical Research, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes